CLINICAL TRIAL: NCT01136538
Title: An Open Label, Balanced, Randomized, Two Treatment, Two-sequence, Two-period, Single-dose Crossover Comparative Bioavailability Study of 1000 mg Valacyclovir HCl Tablets of Dr. Reddys's and Valtrex (R) 1 gm Caplets of GlaxoSmithkline in Healthy Volunteers Under Fed Conditions.
Brief Title: Bioavailability Study of Valacycovir HCl Tablets, 1000 mg of Dr. Reddy's Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. Indu Bhushan/Senior Director, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-VIN-028
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Valacyclovir Hydrochloride
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valacyclovir Hydrochloride (Experimental): Valacyclovir Hydrochloride Tablets, 1000 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Valacyclovir Hydrochloride
- Valtrex (R) (Active Comparator): Valtrex (R) (Valacyclovir Hydrochloride) CAPLETS 1 gram of GlaxoSmithkline
  Interventions: Drug: Valacyclovir Hydrochloride

INTERVENTIONS:
Drug: Valacyclovir Hydrochloride — Valacyclovir Hydrochloride Tablets, 1000 mg of Dr. Reddy's Laboratories Limited
  Other Names: Valtrex (R)(Valacyclovir Hydrochloride) CAPLETS 1 gm

SUMMARY:
The purpose of this study is to

1. Compare and evaluate the single-dose bioavailability study of 1000mg Valacyclovir HCl tablets of Dr. Reddy's and Valtrex (R)(Valacyclovir Hydrochloride)CAPLETS 1 gram of GlaxoSmithkline, in healthy, adult human subjects under fed conditions.
2. monitor the adverse events and ensure the safety of subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-sequence two-period, single-dose, crossover comparative bioavailability study of 1000 mg Valacyclovir Hydrochloride Tablets of Dr. Reddy's Laboratories Ltd., India and valtrex (R) (Valacyclovir Hydrochloride) CAPLETS 1 gram of GlaxoSmithkline in healthy, adult human subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

The subjects were selected for study participation, based on the following criteria:

1. Human subjects aged between 18 and 45 years (including both).
2. Subjects' weight within the normal range according to normal values for the Body Mass Index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable normal range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (PIA view).
6. Have a negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Have negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

The subjects were excluded from the study, based on the following criteria:

1. Hypersensitivity to Valacyclovir Hydrochloride or related drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. History or presence of significant alcoholism or drug abuse in the past one year.
4. History or presence of significant smoking (more than 10 cigarettes or beedi' s/day).
5. History or presence of significant asthma, urticaria or other allergic reactions.
6. History or presence of significant gastric and/or duodenal ulceration.
7. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumour.
8. History or presence of cancer.
9. Difficulty with donating blood.
10. Difficulty in swallowing solids like tablets or capsules.
11. Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg.
12. Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
13. Pulse rate less than 50/minute or more than 100/minute.
14. Oral temperature less than 95°F or more than 98.6°F.
15. Respiratory rate less than 12/minute or more than 20/minute
16. Subjects who have used any prescription medication, within 14 days of period 01 dosing or OTC medication within 14 days of period 01 dosing.
17. Major illness during 3 months before screening.
18. Participation in a drug research study within past 3 months.
19. Donation of blood in the past 3 months before screening.
20. Subjects who have consumed xanthine-containing products (including caffeine, theobromines, etc.) within 48 hours prior to period 01 dosing.
21. Subjects who have consumed food or beverages containing grapefruit or pomelo within 14 days prior to period 01 dosing.
22. Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
23. Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2007-02; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dharmesh Domadia, MD, Principal Investigator — Veeda clinical research Pvt. Ltd., India
Locations (1):
- Veeda clinical research Pvt. Ltd., India, Ahmedabad, Gujarat, India